CLINICAL TRIAL: NCT01884584
Title: Assessment of Potential Use of Indocyanine Green as a Fluorescent Agent for Definition of Surgical Margins in Cancer
Brief Title: Potential Use of Indocyanine Green as a Fluorescent Agent for Definition of Surgical Margins in Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, David A Kooby, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00053609; RAD2162-11 (Other: Other)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Indocyanine green (ICG) (Experimental): ICG will be administered by intravenous infusion over a 20 second period in a 2-8 hour time window before the time of completion of the surgical procedure.
  Interventions: Drug: Indocyanine green (ICG)

INTERVENTIONS:
Drug: Indocyanine green (ICG) — Initial dose of 0.22 mg/kg, which has proven successful in identifying tumor tissue in canine experiments, will be used. The dose will be based on actual body weight. This dose is approximately 40% of the standard human dose for determining cardiac output.
  Other Names: Cardiogreen

SUMMARY:
The surgeon may remove a very small amount of additional tissue compared to what would be removed if you were not enrolled in the study. This tissue may prove to contain tumor or it may contain normal tissue. The surgical cavity will be examined by a special laser pen after the tumor is removed, and if areas of fluorescence are seen, that may indicate tumor cells where the ICG dye collected are still remaining and the surgeon would then remove those. After the tumor and the tissue around it are removed and sent to the laboratory, the tissue may be examined using that same laser pen to see where the cancer cells are and compare that to what the laboratory sees when it looks at the tumor and tissue with a microscope. It is hoped that what the dye shows and what is seen with the microscope will be alike.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To validate the use of intraoperative indocyanine green (ICG) for better definition of tumor margins therefore, minimizing the necessity of a second surgical procedure to obtain negative margins.

OUTLINE:

Patients receive indocyanine green solution intravenously (IV) between 2-8 hours before surgery. Fluorescence measurements are taken from all specimens removed during surgery.

After completion of study, patients are followed up at 48 hours.

ELIGIBILITY:
Inclusion Criteria: Patients with a tumor that will be treated surgically.

Exclusion Criteria:

* Patients with a known history of reaction to iodine or iodine-containing compounds.
* Pregnant women. Any patients found to be pregnant will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The contrast ratio (CR, defined as the integrated fluorescence intensity measured in a known tumor area divided by the integrated fluorescence intensity of a known "not tumor" area) | 1-2 weeks
  Examine the resected tissue to determine whether ICG is sensitive to tumor detection (i.e., whether ICG accumulates in tumor) and whether ICG is specific for tumor (i.e., whether ICG accumulates in normal tissue).

CONTACTS AND LOCATIONS:
Overall Officials: David Kooby, MD, Principal Investigator — Emory University-Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia